CLINICAL TRIAL: NCT01691677
Title: Multicentre, Randomized, Double-blind, Parallel Group, Placebo-Controlled Study on the Therapeutic Efficacy and Safety of Beclomethasone Dipropionate Suspension for Inhalation 800 µg Twice Daily vs. Placebo Added to Antibiotic Therapy in Patients With Acute Rhinosinusitis
Brief Title: beCLomethasone Efficacy in Acute Rhinosinusitis - CLEAR Study
Acronym: CLEAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MC/PR/1400/007/11
Record Dates: First submitted 2012-08-01; First posted 2012-09-25 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Acute Rhinosinusitis
MeSH Terms: interventions — Beclomethasone; Suspensions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- beclomethasone dipropionate (Experimental): beclomethasone dipropionate 800 mcg/2 ml suspension for nebulization,one administration b.i.d. for 14 days
  Interventions: Drug: beclomethasone dipropionate 800 mcg/2 ml suspension for nebulization,one administration b.i.d. for 14 days
- placebo (Placebo Comparator): placebo 2 ml suspension for nebulization, one administration b.i.d. for 14 days
  Interventions: Drug: placebo 2 ml suspension for nebulization, one administration b.i.d. for 14 days

INTERVENTIONS:
Drug: beclomethasone dipropionate 800 mcg/2 ml suspension for nebulization,one administration b.i.d. for 14 days
  Arms: beclomethasone dipropionate
Drug: placebo 2 ml suspension for nebulization, one administration b.i.d. for 14 days
  Arms: placebo

SUMMARY:
Intranasal corticosteroids are beneficial in the treatment of acute rhinosinusitis. As adjunctive therapy to oral antibiotic treatment, mometasone furoate at doses of 200 μg or 400 μg twice daily, was well tolerated and significantly more effective in reducing the symptoms of rhinosinusitis than antibiotic therapy alone. Furthermore,the addition of fluticasone propionate to xylometazoline and antimicrobial therapy with cefuroxime improved clinical success rates and accelerated recovery of patients with a history of chronic rhinitis or recurrent sinusitis who present for treatment of acute rhinosinusitis.

The present study was planned to assess the effects of nebulised beclomethasone dipropionate given as add-on therapy to standard care (oral antibiotics) in the treatment of acute symptomatic rhinosinusitis. Antibiotic therapy will be at the physicians' discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study-related procedures
2. Male and female out-patients aged between 18 and 65 years (inclusive).
3. History of previously diagnosed recurrent or chronic sinusitis that necessitate antibiotic therapy as judged by the investigator.
4. Clinical diagnosis of acute rhinosinusitis defined, according to the European Position Paper on Rhinosinusitis and Nasal Polyps 2007 (20), as the sudden onset of two or more relevant symptoms for <12 weeks, at least one of which is:

   * Nasal blockage/obstruction/congestion, OR
   * Nasal discharge (anterior/posterior nasal drip);

   AND the second one is:

   • Facial pain/pressure or/and reduction/loss of sense of smell.
5. A cooperative attitude and ability to be trained to use correctly the nebuliser with intranasal nose piece.

Exclusion Criteria:

1. Previous sinus surgery;
2. Sinus lavage within the past 7 days;
3. Nasal polyposis or important nasal septum deviation;
4. Antibiotic use (by any route) in the past 30 days;
5. Recurrent moderate epistaxis;
6. Chronic bacterial sinusitis with evidence of failure of antimicrobial therapy;
7. Intranasal or systemic use of corticosteroids within the past 30 days;
8. Chronic use of corticosteroids or immunosuppressive agents;
9. Immunocompromised states;
10. Diagnosis of bronchial asthma or chronic obstructive pulmonary disease (COPD);
11. History of clinically significant cardiac (i.e. congestive heart failure or severe hypertension), renal (i.e. kidney failure), psychiatric (i.e. depression or mood disorders), hepatic (i.e. cholestatic jaundice or hepatic dysfunction), endocrine (i.e. hyperthyroidism or adrenal suppression) or pulmonary disease, or laboratory testing abnormalities, whose sequelae and/or treatments can interfere with the results or treatments of the present study;
12. History of psychiatric diseases likely to require treatment with antidepressant drugs during the study period or treatment with antidepressant drugs in the past 2 weeks;
13. Diagnosis of glaucoma or prostatic hypertrophy;
14. History of alcohol or drug abuse;
15. Allergy, sensitivity or intolerance to study drugs and/or study drugs formulations ingredients (e.g. corticosteroids);
16. Pregnant or lactating women or all women physiologically capable of becoming pregnant UNLESS they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/mL or are using one or more of the following acceptable methods of contraception. surgical sterilization (e.g. bilateral tubal ligation, hysterectomy) hormonal contraception (implantable, patch, oral) double-barrier methods (any double combination of: IUD, male or female condom with spermicidal gel, diaphragm, sponge, cervical cap). A pregnancy test (urine) will be performed at screening in women of childbearing potential.
17. Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study.
18. Participation in another trial in the past 12 weeks or patients previously enrolled in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
proportion of patients who will experience clinical success | 28 days

SECONDARY OUTCOMES:
overall sinus symptoms | 7,14,21,28 days
changes of each symptom | 7, 14, 21, 28 days
level of work performance based on patient perception (recorded on a VAS scale of the diary card) and on missed working time | 7, 14 days
absence of relapses | 7, 14, 21, 28 days
nasal mucociliary transport time | 7, 14 days
nasal air flow resistance | 7, 14 days
Adverse events and adverse drug reactions | 0, 7, 14, 21, 28 days
vital signs | 0, 7, 14, 21, 28 days

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Policlinico Santa Maria alle Scotte, Siena, Italy
  - Ospedale Cisanello, Pisa
  - Policlinico Univesitario Gemelli, Roma

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2011-001459-35